CLINICAL TRIAL: NCT01900223
Title: Chronic Pain After Shoulder Arthroplasty: Epidemiology and Risk Factors.
Brief Title: Chronic Pain After Shoulder Arthroplasty
Status: Completed | Type: Observational
Sponsor: Karen Bjørnholdt (Other)
Collaborators: Central Denmark Region (Other); Augustinus Fonden (Other); Horsens Hospital (Other)
Responsible Party: Sponsor-Investigator, Karen Bjørnholdt, M.D., Ph.D.-student, University of Aarhus
Organization: University of Aarhus (Other)
Other Study IDs: KTB-003
Record Dates: First submitted 2013-07-08; First posted 2013-07-16 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Shoulder prosthesis bearer

SUMMARY:
Chronic pain is relatively common after different types of surgery. The investigators intend to study prevalence, characteristics and risk factors of chronic pain after shoulder arthroplasty, focusing on neuropathic pain characteristics, and risk factors such as preoperative pain, severe acute postoperative pain, age, gender, and pain elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated with any shoulder prosthesis between april 2011 and april 2012 in Denmark

Exclusion Criteria:

* Secondary prosthesis
* Bilateral prosthesis
* Age below 18
* Reoperated in the same shoulder after the prosthesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the Danish Shoulder Arthroplasty Register
Sampling Method: Non-Probability Sample
Enrollment: 786 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Current pain intensity | At time of completing the questionnaire, which is sent to patients 1-2 years after their shoulderprosthesis.
  Pain score by Numeric Rating Scale 0-10

SECONDARY OUTCOMES:
preoperative pain intensity | recalled
  Pain intensity by Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Karen T Bjørnholdt, M.D., Principal Investigator — Aarhus University, Horsens Hospital; Birgitte Brandsborg, M.D., Ph.D., Study Chair — Aarhus University Hospital; Lone Nikolajsen, M.D., DMSc, Study Chair — Aarhus University Hospital; Kjeld Søballe, M.D., DMSc, Study Chair — Aarhus University Hospital